CLINICAL TRIAL: NCT00004127
Title: A Phase II Study of Oxaliplatin in Combination With Fluorouracil and Leucovorin in Carcinoma of the Esophagus and Gastric Cardia
Brief Title: Oxaliplatin Combined With Fluorouracil and Leucovorin in Treating Patients With Recurrent or Metastatic Cancer of the Esophagus or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10015; UCCRC-10015; NCI-T99-0010
Record Dates: First submitted 1999-12-10; First posted 2003-05-07 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Oxaliplatin (85 mg/m2, day 1 of every 14 day cycle), Leucovorin (500 mg/m2, day 1 and 2 of every 14 day cycle), Fluorouracil (Bolus of 400 mg/m2 followed by 22 hr continuous infusion of 600 mg/m2 on days 1 and 2 of every 14 day cycle)
  Interventions: Drug: FOLFOX regimen; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining oxaliplatin with fluorouracil and leucovorin in treating patients who have recurrent or metastatic cancer of the esophagus or stomach.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in patients with recurrent or metastatic carcinoma of the esophagus or gastric cardia receiving the combination of oxaliplatin, fluorouracil, and leucovorin calcium. II. Determine the duration of response and overall survival of this patient population receiving this regimen. III. Determine the toxicity, including neurotoxicity, of this regimen in this patient population.

OUTLINE: This is an open-label, multicenter study. Patients receive oxaliplatin IV over 2 hours on day 1, then leucovorin calcium IV over 2 hours with fluorouracil IV bolus, followed by fluorouracil IV over 22 hours on days 1 and 2. Treatment continues every 2 weeks for a minimum of 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease receive at least 3 additional courses of therapy. Patients are followed for a minimum of 2 years or until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed carcinoma of the esophagus or gastric cardia Stage IV or recurrent Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 10 g/dL Hepatic: Bilirubin normal SGOT less than 2 times upper limit of normal (ULN) Renal: BUN less than 1.5 times ULN Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No congestive heart failure No unstable angina pectoris No myocardial infarction within the past 6 months Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 6 months after study No allergy to platinum compounds or antiemetics appropriate for study No uncontrolled concurrent illness No active infection No clinical evidence of peripheral neuropathy by physical exam or history

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony-stimulating factors during the first course of study Chemotherapy: More than 4 weeks since prior chemotherapy No more than 1 prior chemotherapy regimen for carcinoma of the esophagus or gastric cardia No prior fluorouracil Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified Other: No other concurrent investigational agents No concurrent antiretroviral therapy in HIV-positive patients No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-02; Primary Completion 2002-10 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Mauer, MD, Study Chair — University of Chicago
Locations (22):
- United States (21):
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Columbia LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grant/Riverside Methodist Hospitals, Columbus, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico